CLINICAL TRIAL: NCT07117383
Title: A Phase 1 Pharmacokinetic Study Comparing Hezkue® (ASP-001), Hezkue Turbo® (ASP-001.1), and Select Commercially Available Sildenafil Products Under Fed Conditions in Healthy Adult Male Subjects
Brief Title: Hezkue®, Hezkue Turbo®, and Commercial Sildenafil Products in Fed Healthy Male Subject
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aspargo Labs, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ASP-012-SIL
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-08

CONDITIONS: Erectile Dysfunction
Keywords: erectile dysfunction; Viagra; sildenafil; tadalafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hezkue Formulations (Experimental): Participants in this arm receive a single dose of 100mg (miligrams) of either Hezkue® (ASP-001) or Hezkue Turbo® (ASP-001.1), both liquid formulations containing sildenafil citrate.
  Interventions: Device: ASP-001.1; Drug: ASP-001
- Commercially Available Sildenafil Products (Experimental): Participants in this arm receive a single dose of one of several comparator products, including commercially available sildenafil tablets or sildenafil + tadalafil combination chewables.
  Interventions: Drug: Commercial Sildenafil and Sildenafil/Tadalafil Products

INTERVENTIONS:
Device: ASP-001.1 — Bottle/pump containing ASP-001.1 suspension
  Other Names: Hezkue®, sildenafil citrate oral suspension, sildenafil
  Arms: Hezkue Formulations
Drug: ASP-001 — Oral liquid suspension of sildenafil
  Other Names: Hezkue Turbo®, sildenafil citrate oral suspension, sildenafil
  Arms: Hezkue Formulations
Drug: Commercial Sildenafil and Sildenafil/Tadalafil Products — A selection of marketed sildenafil or sildenafil + tadalafil products used as comparators. Includes tablets and chewables such as Viagra®, Galotam, BlueChew, Aristo Sildaristo, Lemonaid Viagra, Ro Sparks, Hims Hard Mints, and Hello Cake ED Cake Meds.
  Other Names: Viagra®, Galotam, BlueChew, Aristo Sildaristo, Lemonaid Viagra, Ro Sparks, Hims Hard Mints, Hello Cake ED Cake Meds
  Arms: Commercially Available Sildenafil Products

SUMMARY:
The goal of this clinical trial is to compare how different sildenafil formulations are absorbed and tolerated in healthy adult males under fed conditions. The main questions it aims to answer are:

Do Hezkue and Hezkue Turbo differ in absorption compared to other commercial sildenafil products?

Are there any differences in safety or tolerability between the products?

Researchers will compare multiple formulations to evaluate differences in drug absorption and side effects.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn how different formulations of sildenafil-used to treat erectile dysfunction-are absorbed in the body when taken with food, and to understand how safe and well-tolerated they are in healthy adult males. The main questions it aims to answer are:

How do the blood levels of sildenafil compare between Hezkue, Hezkue Turbo, and other commercial sildenafil products?

Do differences in formulation (such as particle size or combination with tadalafil) affect the absorption or safety profile?

Researchers will compare Hezkue and Hezkue Turbo to other sildenafil-containing products (such as Pfizer Viagra, BlueChew, and Ro Sparks) to see if there are differences in how quickly and how much of the drug enters the bloodstream.

Participants will:

* Take a single oral dose of one of the test products after eating a high-fat meal.
* Have blood samples taken over a 4-hour period to measure drug levels.
* Be monitored for side effects and overall health for up to 4 days after each dose.
* Have the option to return for additional visits to test other products, with a 4-day break in between.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be informed of the nature of the study and voluntarily agree to participate by signing an informed consent form prior to any study-specific procedures.
* Participant must be a healthy male, aged 18 to 70 years (inclusive) at the time of dosing.
* Participant must be judged by the Investigator or designee to be in good general health, as documented by medical history, physical examination, clinical laboratory tests, vital signs, and 12-lead electrocardiogram (ECG). Any deviations from normal ranges must be assessed and deemed not clinically significant by the Investigator or designee.
* Participant must have a creatinine clearance (CrCl) value greater than 80 mL/min, as calculated by the Cockcroft-Gault equation.
* Participant must agree to practice an acceptable method of contraception throughout the clinical trial, as outlined in the protocol.

Exclusion Criteria:

* Unwilling or unable to comply with study procedures.
* Use of any investigational drug (except Hezkue/Hezkue Turbo) within 30 days prior to dosing.
* History of significant renal, hepatic, cardiovascular (including orthostatic hypotension), psychiatric, neoplastic, infectious disease, or diabetes mellitus.
* Clinically significant abnormal lab results, vital signs, or ECGs.
* Any hepatic impairment or abnormal liver function tests.
* Positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
* Clinically significant illness within 28 days prior to dosing.
* Known hypersensitivity to sildenafil, tadalafil, vardenafil, or any component of the investigational product (e.g., peppermint oil).
* History of significant food or drug allergies.
* History of drug abuse within the past year or positive drug screen at screening.
* Regular alcohol consumption exceeding 15 units per week.
* Use of CYP450 enzyme inhibitors within 14 days prior to dosing.
* Use of CYP450 enzyme inducers or St. John's Wort within 28 days prior to dosing.
* Blood donation or significant blood loss within 3 months before screening.
* Plasma donation within 14 days prior to first dose.
* Inadequate venous access for repeated blood sampling.
* Difficulty fasting or inability to consume standardized meals.
* Intolerance to fatty foods or inability to consume a high-fat, high-calorie breakfast.
* Difficulty swallowing.
* Regular use of tobacco or nicotine products within 4 weeks prior to screening.
* Major surgery within 3 months or minor surgery within 1 month before screening.
* Considered unsuitable for study participation by the Investigator.
* Institutionalized status.
* Use of hormone replacement therapy within 6 months prior to dosing.
* Consumption of Seville oranges, grapefruit, or pomelo within 7 days prior to dosing.
* Consumption of caffeine, xanthine-containing products, or poppy seeds within 48 hours prior to dosing.
* Receipt of a COVID-19 vaccine within 3 days prior to dosing.
* Presence of braces, retainers, dentures, partial dentures, or tongue piercings.
* Use of nitric oxide donors, organic nitrates/nitrites, antihypertensive medications, or PDE5 inhibitors within 14 days of dosing.
* Blood pressure or heart rate outside acceptable ranges:

  * Systolic BP <90 or >140 mmHg
  * Diastolic BP <50 or >90 mmHg
  * Heart rate <50 or >100 bpm

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Tmax - Time to Maximum Observed Plasma Concentration of Sildenafil | Baseline and up to 4 hours post-dose at 23 specified timepoints
  Measurement of the time (Tmax) to reach maximum observed plasma concentration of sildenafil following a single oral dose under fed conditions.
Cmax - Maximum Observed Plasma Concentration of Sildenafil | Baseline and at 23 timepoints within 4 hours post-dose.
  Measurement of the maximum observed plasma concentration (Cmax) of sildenafil following a single oral dose of study drug.

SECONDARY OUTCOMES:
Number of Participants Reporting Oral Irritation, Dizziness, or Headache | From pre-dose through 96 hours post-dose.
  To assess the frequency and severity of oral irritation, dizziness, or headache following administration of ASP-001.1 (Hezkue Turbo). Descriptive summaries (mean, standard deviation, median, minimum, and maximum) of actual values and changes from baseline will be provided.
Number of Participants With Adverse Events | From pre-dose through 96 hours post-dose.
  The frequency and type of adverse events reported during the study will be summarized, including severity and relationship to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Guralnik, PhD, Principal Investigator — Aspargo Labs, Inc
Locations (1):
- Aspargo Labs, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this study is an early-phase pharmacokinetic trial with a small sample size and limited potential for secondary analyses.